CLINICAL TRIAL: NCT00528736
Title: Plasma B-Type Natriuretic Peptide Concentrations in Preterm Infants < 28 Weeks
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Other Study IDs: EA2/198/05
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Infant, Premature; Ductus Arteriosus, Patent; Natriuretic Peptide Brain
Keywords: preterm infants < 28 weeks; B-type natriuretic peptide; prediction; ductus intervention
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study was to evaluate BNP in preterm infants < 28 weeks on the second day of life, when it is still unknown, if a patent ductus arteriosus is hemodynamic significant or not. We hypothesized that high plasma BNP concentrations on day 2 are associated with the need of PDA intervention in the further course.

DETAILED DESCRIPTION:
From the study infants blood samples (0.1ml) were collected in K-EDTA microtubes within 24 to 48 hours of age through umbilical artery catheter aspiration or routine venous puncture. The samples were spun at 7000 rpm for 3 minutes. Platelet-free plasma was stored at -20°C until BNP analysis of all collected samples was carried out. The BNP assay was performed using a fully automated immunoassay system ADVIA method for the Centaur System (Bayer Diagnostic Division).

In preterm infants who were treated with indomethacin or surgical ligation we collected additional blood samples 2-4 hours before intervention and 24 hours after the completion of the ductus treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written parental informed consent
* Preterm infant < 28 weeks of gestation
* Admitted to our NICU within 48 hours after birth

Exclusion Criteria:

* No written parental informed consent,
* Congenital heart disease,
* Death

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2005-08; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Czernik, MD, Study Director — Department of Neonatology, Charite Virchow Hospital, Medical University Berlin
Locations (1):
- Department of Neonatology, Charite Virchow Hospital, Medical University Berlin, Berlin, State of Berlin, Germany